CLINICAL TRIAL: NCT03867188
Title: The Use of Liposomal Bupivacaine (Exparel) in Soft Tissue Sarcoma Resection
Brief Title: Liposomal Bupivacaine (Exparel) in Sarcomas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment of eligible subjects, delays due to the COVID-19 Virus, and lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00050365; WFBCCC 71118 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-02

CONDITIONS: Soft Tissue Sarcoma; Soft Tissue Tumor; Soft Tissue Tumor and/or Sarcoma
Keywords: Exparel; Liposomal Bupivacaine; Removal by Surgery; Pain Reduction
MeSH Terms: conditions — Sarcoma; Soft Tissue Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liiposomal Bupivacaine Group (Experimental): Qualified participants with a soft tissue sarcoma of the thigh will be given the alternative protocol utilizing liposomal bupivacaine (Exparel®). The alternative protocol will utilize general or spinal anesthesia, but will also include the use of intraoperative liposomal bupivacaine instead of a regional nerve block.
  Interventions: Drug: Liposomal Bupivacaine
- Control Group (No Intervention): A retrospective control group will be assembled from electronic medical records of 3 patients who underwent resection of a soft tissue sarcoma of the thigh and will be accessed and analyzed for the variable of interest.

INTERVENTIONS:
Drug: Liposomal Bupivacaine — A 25 gauge or larger bore needle will be used to inject the liposomal bupivacaine at the site of operation following the prescription guidelines provided by Exparel®. The maximum dose allowable for this study is 266mg or 20 mL as indicated in the FDA package insert.
  Other Names: Exparel
  Arms: Liiposomal Bupivacaine Group

SUMMARY:
The purpose of this research is to study a medication called liposomal bupivacaine (EXPAREL®). Study doctors want to see if it is safe, if it can reduce pain after surgery, and the study doctor want to study its use after the removal a soft tissue tumor called a sarcoma

DETAILED DESCRIPTION:
The hypothesis for this project is that using liposomal bupivacaine will reduce patients' morphine equivalent usage postoperatively while maintaining similar pain scores and lengths of stay when compared to patients that did not receive intraoperative liposomal bupivacaine. Thus, if the use of liposomal bupivacaine proves to aid in pain control and the reduction of initial opiate use following soft tissue sarcoma resection, it could be reasonably suggested that liposomal bupivacaine become incorporated into a multimodal form of pain management following soft tissue sarcoma resection. These results are expected to have a significant positive impact; allowing for a reduction in narcotic pain medication usage and its associated side effects while decreasing health care expenditures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a soft tissue sarcoma of the thigh
* Must have sufficient health to withstand the physical demands of surgery
* ≥ 18 years old
* ECOG performance status of ≤ 2
* Ability to understand and the willingness to sign an IRB-approved informed consent document

Exclusion Criteria:

* History of clinically significant medical conditions including: Cardiovascular: Atrial Fibrillation, Ventricular Fibrillation, Significant Coronary Artery Disease. Hepatic: Viral or Autoimmune Hepatitis, Cirrhosis of the Liver, Liver Metabolism Disorders. Renal: Any form of renal impairment. EXPAREL® is cleared by the kidneys, thus any form of renal impairment could lead to an adverse reaction.
* Medical condition(s) or concurrent surgery that may have required analgesic treatment in the postoperative period for pain that was not strictly related to the study surgery.
* Any clinically significant event or condition discovered during surgery that may have complicated the patient's post surgical course such as vascular or nerve involvement that was unknown before surgery.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to liposomal bupivacaine.
* Pregnant women are excluded from this study because EXPAREL has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EXPAREL, breastfeeding should be discontinued if the mother is treated with EXPAREL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with peak pain scores measured by VAS less than 7 | Up to 24 hours
  Feasibility of Exparel for post surgical pain management in soft-tissue sarcoma surgeries of the thigh will be defined as peak pain score measured by VAS (Visual Analogue Scale) less than 7. VAS scores range 0 (no pain) to 10 (unbearable pain). Higher scores denote worse outcome measures.

SECONDARY OUTCOMES:
Peak Pain Scores during hospital stay post surgery | Up to 5 days
  Peak pain scores will be measured by VAS (Visual Analogue Scale) which is printed on the Post-Operative Pain and Medication Administration questionnaire. VAS ranges 0 (no pain) to 10 (unbearable pain). Higher scores denote worse outcome measures.
Amount of opiate use post-operatively while the patient is in the hospital in milligram morphine equivalent (MME) | Up to 5 days
  The opioid medications that the subject uses will be recorded and the data regarding total narcotic usage will be converted to MME to maintain a standard unit for the study.
Number of surgical-related infection | 6 week post surgery
  Number of surgical-related infection will be documented by use of Treatment Follow-Up Form and Adverse Event Log.
Average Pain Scores during hospitalization | up to 5 days
  Average pain scores will be measured by VAS (Visual Analogue Scale). VAS ranges 0 (no pain) to 10 (unbearable pain). Higher scores denote worse outcome measures.
Length of time in hospital | End of hospitalization (up to 30 days)
  The unit of time used to record length of stay will be days. Defined as the time from entry into the post anesthesia care unit (PACU) to discharge
Rate of approached and consented patients | end of the study up to 2 years
  The rate will be calculated with the number of participants that consented divided by the number of patients approached about the study

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Emory, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication, no end date
Access Criteria: Anyone who wishes to access the data; Any purpose. Data available indefinitely.

REFERENCES:
- [Background] Baxter R, Bramlett K, Onel E, Daniels S. Impact of local administration of liposome bupivacaine for postsurgical analgesia on wound healing: a review of data from ten prospective, controlled clinical studies. Clin Ther. 2013 Mar;35(3):312-320.e5. doi: 10.1016/j.clinthera.2013.02.005. Epub 2013 Mar 1. PMID 23453403
- [Background] Exparel (bupivacaine liposomal) [prescribing information]. San Diego, CA: Pacira Pharmaceuticals Inc; August 2016
- [Background] Ranawat AS, Ranawat CS. Pain management and accelerated rehabilitation for total hip and total knee arthroplasty. J Arthroplasty. 2007 Oct;22(7 Suppl 3):12-5. doi: 10.1016/j.arth.2007.05.040. PMID 17919586
- [Background] Snyder MA, Scheuerman CM, Gregg JL, Ruhnke CJ, Eten K. Improving total knee arthroplasty perioperative pain management using a periarticular injection with bupivacaine liposomal suspension. Arthroplast Today. 2016 Jan 11;2(1):37-42. doi: 10.1016/j.artd.2015.05.005. eCollection 2016 Mar. PMID 28326395
- See also: North Carolina Medical Board. Stop Act prescribing limits in effect January 1, 2018. Accessed January, 30 2018. — https://www.ncmedboard.org/resources-information/professional-resources/publications/forum-newsletter/notice/stop-act-prescribing-limits-in-effect-jan

DOCUMENTS (1):
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03867188/ICF_000.pdf